CLINICAL TRIAL: NCT01879501
Title: Living Successfully With Chronic Eye Diseases: the 'Living Successfully With Low Vision' (LSLV) Program - a Randomized Controlled Trial of a Self-management Program for Low Vision
Brief Title: Living Successfully With Chronic Eye Diseases
Acronym: ADAPT-LAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: Ministry of Health, Singapore (Other Government); University of Melbourne (Other); Singapore National Eye Centre (Other Government); Curtin University (Other)
Responsible Party: Principal Investigator, Peggy Pei-Chia Chiang, Doctor, Singapore Eye Research Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSRG11MAY005
Record Dates: First submitted 2013-04-10; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Diseases; Low Vision; Diabetic Retinopathy; Glaucoma; Age-related Macular Degeneration
Keywords: Low vision; Self management; Randomized controlled trial; Quality of life; Self efficacy; Effectiveness; Chronic eye diseases management
MeSH Terms: conditions — Chronic Disease; Vision, Low; Diabetic Retinopathy; Glaucoma; Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Vision Self-Management Program (Experimental): Intervention: The program will work with participants to choose a specific and achievable goal they wish to achieve, involve participants in the learning process, provide information, explore experiences with low vision, and solutions to develop problem solving skills to enhance self efficacy. Participants will learn new techniques to cope with their activities of daily living. In addition to this, local guest experts in the field will be sourced and invited to provide training in aspects of low vision care.
  Interventions: Behavioral: Low Vision Self-Management Program
- Usual Care (No Intervention): Usual care delivered at the Singapore National Eye Centre

INTERVENTIONS:
Behavioral: Low Vision Self-Management Program — The program has been describe above.
  Arms: Low Vision Self-Management Program

SUMMARY:
The need for low vision services (LVS) will increase exponentially over the coming years due to the anticipated and exponential growth in the ageing population in Singapore and a rise in chronic non-communicable eye diseases. Finding the best evidenced-based management for chronic eye diseases contributing to low vision (LV) is therefore crucial. Improving patient responsibility is the key to managing LV effectively.1 This means achieving optimum self management (SM).2 However, there are currently no LV SM programs in Singapore and none has been evaluated using a randomized controlled trial (RCT) design, the gold standard methods to evaluate health interventions.

The aims of this study are to assess the effectiveness of the 'Living Successfully with Low Vision (LSLV)' program in improving quality of life (QoL) in 160 elderly people with LV attending the Singapore National Eye Centre (SNEC) LV clinic. Of these, 80 will be randomly allocated to receive the LSLV 4-week SM program while the remaining 80 will receive the usual care. Comparisons will be made to determine the efficacy of the LSLV program. QoL, self-efficacy, emotional well being, and vision-specific distress will be assessed 2 weeks after training, and at six months and 12 months post intervention.

This study will be the first evidenced-based RCT investigating the effectiveness of a novel vision-specific self-management strategy to improve QoL. It will also adopt a longitudinal design where the effectiveness of these interventions will be evaluated at 12 months-the first follow-up assessment of that duration at both national and international levels. Furthermore this will be the first study to characterize and profile the patients where the effect of the program did not demonstrate an improvement in both primary and secondary outcomes six months after its completion. The future clinical implications of this study include the potential to implement a successful model of LV rehabilitation in other tertiary centres around the country.

DETAILED DESCRIPTION:
The need for low vision services (LVS) will increase exponentially over the coming years due to the anticipated and exponential growth in the ageing population in Singapore and a rise in chronic non-communicable eye diseases. Finding the best evidenced-based management for chronic eye diseases contributing to low vision (LV) is therefore crucial. Improving patient responsibility is the key to managing LV effectively.1 This means achieving optimum self management (SM).2 However, there are currently no LV SM programs in Singapore and none has been evaluated using a randomized controlled trial (RCT) design, the gold standard methods to evaluate health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years to 75 years
* Visual acuity ≤6/12 to ≤6/480 in the better eye after best correction OR
* Visual field of less than 10 degrees from the point of fixation, but with the potential to use vision for the planning and/or execution of a task
* Duration of low vision ≥ 2 years
* No cognitive impairment (as assessed with the 6-item cognitive impairment test)
* Have adequate hearing with/without aids to respond to normal conversation

Exclusion Criteria:

* Not matching the above

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Vision-related quality of life | up to 12 months post intervention

SECONDARY OUTCOMES:
Perceived self-efficacy, emotional well being, and vision-specific distress | baseline (before randomization to either usual care or intervention group); 2 weeks, 6 months and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peggy PC Chiang, PhD, Principal Investigator — Singapore Eye Research Institute (SERI)
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore